CLINICAL TRIAL: NCT00003316
Title: Evaluation of Gemcitabine in the Treatment of Recurrent or Persistent Leiomyosarcoma of the Uterus
Brief Title: Gemcitabine in Treating Patients With Recurrent or Refractory Cancer of the Uterus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000066265; GOG-131E
Record Dates: First submitted 2000-11-06; First posted 2004-04-09 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2004-05

CONDITIONS: Sarcoma
Keywords: recurrent uterine sarcoma; uterine leiomyosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Gemcitabine

INTERVENTIONS:
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine in treating patients with recurrent or refractory cancer of the uterus.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the antitumor activity of gemcitabine in patients with recurrent or persistent leiomyosarcoma of the uterus who failed higher priority treatment protocols. II. Determine the toxicity of gemcitabine in these patients.

OUTLINE: Patients receive gemcitabine IV over 30 minutes weekly for 3 weeks. Courses repeat every 4 weeks in the absence of unacceptable toxicity and disease progression. Patients with partial response, complete response, or stable disease receive at least 3 courses of therapy. Patients are followed every 3 months for 2 years, then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent or persistent uterine leiomyosarcoma that is refractory to curative therapy or standard treatments Failed local therapeutic measures and considered incurable Measurable disease Not eligible for a higher priority GOG protocol

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Granulocyte count at least 1,500/mm3 Hepatic: Bilirubin no greater than 1.5 times normal SGOT no greater than 3 times normal Alkaline phosphatase no greater than 3 times normal Renal: Creatinine no greater than 1.5 mg/dL Other: No significant infection At least 5 years since any other invasive malignancy except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since prior biologic therapy Chemotherapy: At least 3 weeks since prior chemotherapy and recovered No prior gemcitabine No more than 1 prior chemotherapy regimen (single agent or combination therapy) Endocrine therapy: At least 3 weeks since prior endocrine therapy Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Surgery: At least 3 weeks since prior surgery and recovered

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-08; Primary Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Y. Look, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (40):
- United States (39):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Radiation Oncology Branch, Bethesda, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- NCIC-Clinical Trials Group, Kingston, Ontario, Canada

REFERENCES:
- [Result] Look KY, Sandler A, Blessing JA, Lucci JA 3rd, Rose PG; Gynecologic Oncology Group (GOG) Study. Phase II trial of gemcitabine as second-line chemotherapy of uterine leiomyosarcoma: a Gynecologic Oncology Group (GOG) Study. Gynecol Oncol. 2004 Feb;92(2):644-7. doi: 10.1016/j.ygyno.2003.11.023. PMID 14766260